CLINICAL TRIAL: NCT00233519
Title: Effects of SomatoKine (Iplex) (rhIGF-I/rhIGFBP-3) in Myotonic Dystrophy Type 1 (DM1)
Brief Title: Effects of SomatoKine (Iplex)Recombinant Human Insulin-like Growth Factor-1/Recombinant Human Insulin-like Growth Factor-binding Protein-3 (rhIGF-I/rhIGFBP-3) in Myotonic Dystrophy Type 1 (DM1)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Imsmed Incorporated (Industry)
Responsible Party: Principal Investigator, Richard T Moxley, Professor of Neurology, University of Rochester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5 U54 NS048843-03 A; 5U54NS048843-03 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Myotonic Dystrophy
MeSH Terms: conditions — Myotonic Dystrophy | interventions — somatoKine; IGF-I-IGFBP-3 complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1- Two Escalating Doses of Iplex (Experimental): 0.5 and 1.0 mg/kg/day
  Interventions: Drug: SomatoKine/IPLEX
- Cohort 2 - Three Escalating Doses of Iplex (Active Comparator): 0.5, 1.0, and 2.0 mg/kg/day
  Interventions: Drug: SomatoKine/IPLEX

INTERVENTIONS:
Drug: SomatoKine/IPLEX — Cohort 1: self-administered subcuteanous injections of 0.5 mg/kg/day of iPlex for 8 weeks, followed by 1.0 mg/kg/day of iPlex for 16 weeks.
  Cohort 2: consecutive 8 week treatments of 0.5, 1.0, and 2.0 mg/kg/day of iPlex for a total of 24 weeks by self-administered subcuteanous injection.

SUMMARY:
The aim of this study is to investigate the safety and feasibility of daily subcutaneous injections of recombinant IGF1 complexed with IGF binding protein 3 (SomatoKine-INSMED) as a treatment for muscle wasting and weakness in myotonic dystrophy type 1.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of DM-1 according to accepted clinical research criteria.23 The clinical research criteria require each of the following: (1) clinically evident myotonia; (2) muscle weakness in a characteristic distribution (distal predominant); and (3) similar findings in a first degree relative.
* Age 21 to 60 years (inclusive).
* Ability to walk 30 feet without assistance (cane and leg bracing is permitted).
* Weakness of sufficient severity to justify treatment and provide a reasonable opportunity to observe a therapeutic effect. At the eligibility evaluation, eligible patients must show both of the following:

  1. muscle strength in a distal muscle group (ankle dorsiflexors or deep flexors of the fingers) which is less than or equal to grade 4 (Medical Research Council grade).
  2. muscle strength in a proximal or mid-limb muscle group (flexors or extensors of the knee, elbow, shoulder, or hip) which is which is greater than or equal to 4- (Medical Research Council grade).
* For patients that are not within driving distance to Rochester, a local health care provider in their area must be able to complete their home visits.
* Competent, willing, and able to give informed consent.
* Able to self-administer study medication by subcutaneous injection or caregiver available to administer study medication.

Exclusion Criteria:

* Congenital DM-1. Congenital disease constitutes ~10% of all cases of DM-1. Early in life, the weakness in individuals with congenital DM-1 derives from maldevelopment of skeletal muscle rather than muscle degeneration. Later in life, these individuals are also subject to the added effects of a wasting process similar to classical DM-1. However, it is difficult to determine which of these phenomena are mainly to blame for weakness in a particular patient. Furthermore, more than 75% of patients with congenital DM-1 have mental retardation.
* Prior treatment with glucocorticoids, anabolic steroids, testosterone, growth hormone, or IGF-I within 1 year of entry; or any investigational agent within 60 days of entry.
* Any history of malignancy except for surgically cured skin cancer or pilomatricoma (benign tumor of the hair follicle that is associated with DM-1).
* Women of childbearing potential who are not using effective birth control; women who are pregnant or lactating.
* Medical illness which would prevent assessment of muscle strength or function. This exclusion would include individuals with orthopedic, cardiac, or pulmonary disorders which preclude proper positioning on the myometry testing table, or restrict their ability to tolerate repeated maximum muscle contractions.
* Known allergy to tetracycline.
* Diaphragmatic weakness such that patients are unable to tolerate supine position, or swallowing impairment such that patients are unable to maintain nutrition without use of gastrostomy.
* Symptomatic liver or kidney disease, insulin requiring diabetes or type 2 diabetes requiring oral anti-diabetic agents.
* Untreated thyroid disease (hypo or hyperthyroidism)
* Major psychiatric illness (major depression, bipolar disorder, or schizophrenia) within twelve months of entry.
* History of non-compliance with other therapies.
* Drug or alcohol abuse within 12 months of enrollment.
* In men, evidence of a mass lesion on clinical examination by their primary care physician within twelve months prior to entry into the study (specifically prostate or testicular mass on clinical exam or other signs of mass lesion) or evidence of mass lesion on chest x-ray. In men 50 years of age or older, prostate specific antigen (PSA) elevation above normal.
* In women, evidence for mass lesion on clinical examination by their primary care physician or gynecologist (specifically breast & pelvic exam) within 12 months of entry into the study or evidence of mass lesion on chest x-ray. In women 40 years of age or older, evidence of mass lesion on mammogram. Women with Gail Scores > 1.7 will be excluded due to their increased risk of developing cancer.
* Atrial fibrillation/flutter; 2nd or 3rd degree heart block without pacemaker treatment
* Weight greater than 100 kilograms(kg).
* Body Mass Index greater than 30.
* History of bleeding diathesis or use of anticoagulant medications. Patients taking nonsteroidal anti-inflammatory agents will be asked to discontinue these medications 3 days prior to muscle biopsy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Moxley, III, M.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Heatwole CR, Eichinger KJ, Friedman DI, Hilbert JE, Jackson CE, Logigian EL, Martens WB, McDermott MP, Pandya SK, Quinn C, Smirnow AM, Thornton CA, Moxley RT 3rd. Open-label trial of recombinant human insulin-like growth factor 1/recombinant human insulin-like growth factor binding protein 3 in myotonic dystrophy type 1. Arch Neurol. 2011 Jan;68(1):37-44. doi: 10.1001/archneurol.2010.227. Epub 2010 Sep 13. PMID 20837825
- See also: Webpage for the National Registry of Myotonic Dystrophy and Facioscapulohumeral Dystrophy patients and their family members. — http://www.dystrophyregistry.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1- Two Escalating Doses of iPlex: N=6 This group received self-administered subcuteanous injections of 0.5 mg/kg/day of iPlex for 8 weeks, followed by 1.0 mg/kg/day of iPlex for 16 weeks.
- Cohort 2-Three Escalating Doses of iPlex: N=9 Following approval of the safety monitoring committee who reviewed the data on the cohort 1, the second cohort received consecutive 8 week treatments of 0.5, 1.0, and 2.0 mg/kg/day of iPlex for a total of 24 weeks by self-administered subcuteanous injection.
Period: Overall Study
Arm/Group | Cohort 1- Two Escalating Doses of iPlex | Cohort 2-Three Escalating Doses of iPlex
Started | 7 | 10
Completed | 6 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- Two Escalating Doses of iPlex | Cohort 2-Three Escalating Doses of iPlex | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Number of Study Participants Who Safely Tolerated Somatokine
Description: Safety and tolerability was measured via interval laboratory studies,electrocardiograms, echocardiograms, ultrasounds of the abdomen and pelvis, dual energy x-ray absorptiometry (DEXA) studies, chest and neck x-rays, and serial physical examinations. The participants had six inpatient evaluations at the University of Rochester General Clinical Research Center (Weeks 0, 8, 16, 24, 28, and 40) and nine outpatient evaluations. Patients also completed side effects diaries to record any adverse events in the interval time between inpatient and outpatient evaluations.
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Cohort 1- Two Escalating Doses of iPlex | Cohort 2-Three Escalating Doses of iPlex
Number analyzed (Participants) | 6 | 9
participants | 6 | 9

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Cohort 1- Two Escalating Doses of iPlex | Cohort 2-Three Escalating Doses of iPlex
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/9
Other Adverse Events (participants affected / at risk) | 3/6 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- Two Escalating Doses of iPlex (N=6) | Cohort 2-Three Escalating Doses of iPlex (N=9)
Acute Inflammation of Gallbladder (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort 1- Two Escalating Doses of iPlex (N=6) | Cohort 2-Three Escalating Doses of iPlex (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bilateral swelling of optic nerves (Eye disorders) | 0 (0) | 1 (1)
blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 0 (0) | 1 (1)
bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Change in size of moles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0)
Cold sensation in esophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cut on top of head (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cyst left ovary (Reproductive system and breast disorders) | 0/2 (0) | 1/5 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Elevated thyroid stimulating hormone (TSH) level (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Eyelid dysfunction (Eye disorders) | 0 (0) | 1 (1)
Fell on ice, hit left knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Film on both eyes (Eye disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 1 (3)
Gallstone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 1/4 (1) | 0/4 (0)
Halos (Eye disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 2 (2) | 3 (7)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 2 (2)
Hyperkelmia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypovolemia (Vascular disorders) | 0 (0) | 1 (1)
Increase in moles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased need for sleep (General disorders) | 0 (0) | 1 (1)
Increased thirst (General disorders) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Left chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Left knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left pinky pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lump (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mood alteration/depression (Psychiatric disorders) | 0 (0) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Papules (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rubor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin excision (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin tag-moles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small raised red dots (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Twisted ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Upper posterior pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Venostasis (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
National Institutes of Health (NIH) can review the content of planned submissions prior to public release (3 weeks notice requested) to insure integrity of the NIH and the Data Safety Monitoring Board (DMSB)staff.